CLINICAL TRIAL: NCT05304130
Title: A Single Center, Single Dose, Open-label Study in Healthy Japanese Participants to Evaluate the Safety, Tolerability, and Pharmacokinetics of Otilimab
Brief Title: A Study in Healthy Japanese Participants to Evaluate the Safety and Pharmacokinetics of Otilimab
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: This study was cancelled because of the limited efficacy demonstrated in the ContRAst phase III programme as a potential treatment for rheumatoid arthritis. GSK has decided not to progress with regulatory submissions
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 208326
Record Dates: First submitted 2022-03-22; First posted 2022-03-31 (Actual); Last update posted 2023-01-26 (Actual); Status verified 2023-01

CONDITIONS: Arthritis, Rheumatoid
Keywords: Japanese participants; Otilimab; Pharmacokinetics; Rheumatoid arthritis; Safety; Tolerability
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — Otilimab

STUDY DESIGN:
Intervention Model Description: Eligible participants will receive treatment with otilimab.
Masking Description: This is an open-label study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Healthy Japanese participants receiving otilimab (Experimental)
  Interventions: Biological: Otilimab

INTERVENTIONS:
Biological: Otilimab — Otilimab will be administered via pre-filled syringe.

SUMMARY:
This study will assess the safety, tolerability and pharmacokinetics (PK) profiles of otilimab in healthy Japanese participants.

ELIGIBILITY:
Inclusion criteria:

* Participant must be 20 to 50 years of age inclusive, at the time of signing the informed consent.
* Japanese participants who are overtly healthy as determined by medical evaluation including medical history, physical examination, laboratory tests, and cardiac monitoring.
* A Coronavirus Disease-2019 (COVID-19) screening with negative test: Two consecutive approved molecular tests (Polymerase chain reaction [PCR] or antigen test) separated by greater than (>)24 hours. The second test should be within 72 hours of admission to the unit on Day -1.
* Body mass index (BMI) within the range 18.5 to 24.9 kilograms per meter square (kg/m^2) (inclusive).

Exclusion Criteria:

* History or presence of cardiovascular, respiratory, hepatic, renal, gastrointestinal, endocrine, hematological, or neurological disorders capable of significantly altering the absorption, metabolism, or elimination of drugs; constituting a risk when taking the study treatment; or interfering with the interpretation of data.
* Active infections (including localized infections), or history of recurrent infections (excluding recurrent fungal infections of the nail bed), or has required management of acute or chronic infections
* History of any respiratory disease which (in the opinion of the investigator) would compromise participant safety or the ability of the participant to complete the study.
* Clinically-significant or unstable (in the opinion of the investigator) persistent cough or dyspnea that is unexplained.
* Current or previous active Tuberculosis (TB), history of untreated or incompletely treated active or latent TB, suspected or known extra pulmonary TB.
* Previous close contact with a person with active TB and did not receive satisfactory anti-tuberculosis treatment as per World Health Organization (WHO) or national guidelines.
* Hemoglobin less than or equal to (<=)9 grams per deciliter (g/dL); white blood cell (WBC) count <=3.0 times 10^9/ Liter (L); platelet count <=100 times 10^9/L; absolute neutrophil count (ANC) <=1.0 times 10^9/L; lymphocyte count <=0.75 times 10^9/L at screening.
* A vaccination (live or attenuated) within 30 days prior to Day 1 or Bacillus Calmette-Guerin (BCG) vaccination within 365 days prior to Day 1, or a live vaccination planned during the course of the study. Any COVID-19 vaccination within 14 days prior to enrolment.
* Any surgical procedure, including bone or joint surgery/synovectomy within 8 weeks prior to Day 1 or any planned surgery within the duration of the study.
* Significant allergies to humanized Monoclonal antibody (mAb).
* Participants with known COVID-19 positive contacts within 14 days prior to screening.
* History of lymphoma, leukemia, or any malignancy.
* History of infected joint prosthesis at any time, with the prosthesis still in situ. History of leg ulcers, catheters, chronic sinusitis or recurrent chest or urinary tract infections.
* Use of prescription or non-prescription drugs within 7 days (or 14 days if the drug is a potential enzyme inducer) or 5 half-lives (whichever is longer) before the start of study intervention until completion of the evaluation visit, unless, in the opinion of the investigator and sponsor, the medication will not interfere with the study.
* Treatment with biologic agents (such as mAb including marketed drugs) within 3 months or 5 half-lives (whichever is longer) prior to dosing.
* Blood donation/sampling within 60 days prior to screening.
* The participant with positive Serological test for syphilis, Human immunodeficiency virus (HIV) antigen/antibody, or Human T-cell lymphotropic virus type 1 (HTLV-1) antibody.
* The participant with positive test for Hepatitis B surface antigen (HBsAg), Hepatitis B core antibody (HBcAb), Hepatitis B surface antibody (HBsAb), or Hepatitis C virus (HCV) antibody.
* Positive pre-study drug/alcohol screen.
* Participants with signs and symptoms suggestive of COVID-19 (fever, cough) within 14 days prior inpatient admission on Day -1.

Ages: 20 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2023-02-08 (Estimated); Primary Completion 2023-05-04 (Estimated); Study Completion 2023-05-04 (Estimated)

PRIMARY OUTCOMES:
Maximum drug concentration (Cmax) following administration of otilimab | Up to 8 Weeks
Area under the concentration-time curve from pre-dose to infinity (AUC[0-infinity]) following administration of otilimab | Up to 8 Weeks

SECONDARY OUTCOMES:
Area under the plasma concentration-time curve from pre-dose to t (AUC[0-t]) following administration of otilimab | Up to 8 Weeks
Time to maximum plasma concentration (Tmax) following administration of otilimab | Up to 8 Weeks
Elimination half-life (t1/2) following administration of otilimab | Up to 8 Weeks
Time to reach the last quantifiable plasma concentration (Tlast) following administration of otilimab | Up to 8 Weeks
Number of participants with Adverse events (AEs), Serious adverse events (SAEs) and Adverse events of special interests (AESIs) | Up to 8 weeks
Change from Baseline in hematology parameters: Basophils, Eosinophils, Lymphocytes, Monocytes, Neutrophils and Platelet count (Giga cells per liter) | Baseline and up to 8 weeks
Change from Baseline in hematology parameter: Red blood cell (RBC) count (Trillion cells per liter) | Baseline and up to 8 weeks
Change from Baseline in hematology parameter: Hemoglobin (Grams per Liter) | Baseline and up to 8 weeks
Change from Baseline in hematology parameter: Hematocrit (Proportion of red blood cells in blood) | Baseline and up to 8 weeks
Change from Baseline in hematology parameter: Mean Corpuscular Volume (MCV) (Femtoliters) | Baseline and up to 8 weeks
Change from Baseline in hematology parameter: Mean corpuscular hemoglobin (MCH) (Picograms) | Baseline and up to 8 weeks
Change from Baseline in hematology parameter: Percentage of reticulocytes (Percentage of reticulocytes) | Baseline and up to 8 weeks
Change from Baseline in clinical chemistry parameters: Alanine aminotransferase (ALT), Alkaline phosphatase (ALP), Aspartate aminotransferase (AST), Creatine kinase, Gamma Glutamyl transferase (GGT), Lactate Dehydrogenase (International units per Liter) | Baseline and up to 8 weeks
Change from Baseline in clinical chemistry parameters: Calcium, glucose, potassium, sodium, Chloride, Phosphate and Blood urea nitrogen (BUN) (Millimoles per Liter) | Baseline and up to 8 weeks
Change from Baseline in clinical chemistry parameters: Creatinine, direct bilirubin, total bilirubin and uric acid (Micromoles per liter) | Baseline and up to 8 weeks
Change from Baseline in clinical chemistry parameters: Albumin and Total protein (Grams per liter) | Baseline and up to 8 weeks
Change from Baseline in clinical chemistry parameter: C-reactive protein (CRP) (Milligrams per liter | Baseline and up to 8 weeks
Change from Baseline in clinical chemistry parameter: Amylase (Units per liter) | Baseline and up to 8 weeks
Change from Baseline in lipid panel parameters: Total cholesterol, low-density lipoprotein (LDL) cholesterol, high-density lipoprotein (HDL) cholesterol and triglycerides (Millimoles per Liter) | Baseline and up to 8 weeks
Number of participants with abnormal urinalysis parameters by Dipstick Method | Baseline and up to 8 weeks
Change from Baseline in vital signs: Systolic Blood Pressure (SBP) and Diastolic Blood Pressure (DBP) (Millimeters of mercury) | Baseline and up to 8 weeks
Change from Baseline in vital sign: Pulse rate (Beats per minute) | Baseline and up to 8 weeks
Change from Baseline in vital signs: Body temperature (Degrees Celsius) | Baseline and up to 8 weeks
Change from Baseline in Electrocardiogram (ECG) parameters: PR interval, QRS duration, QT interval and corrected QT (QTc) interval (Milliseconds) | Baseline and up to 8 weeks
Number of participants with anti-drug antibodies (ADAs) to otilimab | Up to Week 8
Number of participants with drug-neutralizing antibodies to otilimab | Up to Week 8

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline

IPD SHARING:
Plan to Share IPD: Yes
IPD for this study will be made available via the Clinical Study Data Request site.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: IPD will be made available within 6 months of publishing the results of the primary endpoints, a key secondary endpoints and safety data of the study.
Access Criteria: Access is provided after a research proposal is submitted and has received approval from the Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months but an extension can be granted, when justified, for up to another 12 months.
URL: http://clinicalstudydatarequest.com